CLINICAL TRIAL: NCT01786434
Title: Routine Versus on Demand Administration of Fentanyl in Colonoscopy: A Multi-centre Randomized Controlled Trial
Brief Title: Routine or On-demand Fentanyl in Colonoscopy
Acronym: FEKOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/1737
Record Dates: First submitted 2013-01-03; First posted 2013-02-08 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Pain
Keywords: colonoscopy; pain
MeSH Terms: conditions — Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine medication arm (Experimental): Fentanyl is given routinely to all patients before the procedure
  Interventions: Drug: Routine medication arm
- Fentanyl on-demand arm (Active Comparator): Fentanyl is given during the procedure if the patient experiences pain
  Interventions: Drug: Fentanyl on-demand arm

INTERVENTIONS:
Drug: Routine medication arm — 50 micrograms of fentanyl given before the procedure
  Other Names: fentanyl
  Arms: Routine medication arm
Drug: Fentanyl on-demand arm — Fentanyl 50 microgram is provided on-demand, that is, if the patient has pain during the procedure.
  Other Names: Fentanyl
  Arms: Fentanyl on-demand arm

SUMMARY:
Colonoscopy may be an unpleasant procedure. Sedation and/or analgesics is therefore routinely administered in most countries. In Norway, however, routine sedation is rare, and medication is normally given on demand, that is, if necessary during the procedure. The investigators want to evaluate whether the effect of fentanyl, a synthetic opioid with fast onset of action, is better given before the procedure than during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Referred for out-patient colonoscopy

Exclusion Criteria:

* ASA-score 3 or higher
* Same day upper endoscopy
* Pregnancy
* Pacemaker
* Patient require medication before colonoscopy
* Previous resection of colon or rectum
* Significant psychiatric morbidity
* Oxygen saturation < 95% without supplementary oxygen
* Contra indications to fentanyl
* Inability to sign inform consent
* Inability to understand information about the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Pain during colonoscopy | Immediately after the procedure and after 24 hours
  Pain is recorded on a 4 point Likert scale and a 100 mm VAS scale.

SECONDARY OUTCOMES:
Additional medication | During the colonoscopy
  The investigators want to assess the need for additional medication during the colonoscopy in the "routine fentanyl-arm" compared to the "fentanyl on-demand arm".

OTHER OUTCOMES:
Patient satisfaction | The day after the procedure
  Patients are asked about satisfaction with information and treatment (yes/no)
Complications | During the procedure
  Sedation-related complications during the procedure
Caecum intubation time | During the procedure
  Time to reach the caecum (minutes)
Caecum intubation rate | During the procedure
  The number of complete procedures divided by the total number of procedures
Willingness to repeat | Within one hour after the procedure
  The patient is asked whether he/she would be willing to have the procedure again in the same way (yes/no).
Recovery time | Immediately after the procedure Within one hour after the procedure
  Time elapsing between end of procedure until leaving the department

CONTACTS AND LOCATIONS:
Overall Officials: Oyvind Holme, MD, Principal Investigator — Sorlandet Hospital HF
Locations (1):
- Sorlandet Hospital Kristiansand, Kristiansand, Norway

REFERENCES:
- [Derived] Holme O, de Lange T, Stallemo A, Wiig H, Hasund A, Dvergsnes K, Garborg K, Ystrom CM, Loberg M, Hoff G, Bretthauer M, Kalager M. Routine vs. on-demand analgesia in colonoscopy: a randomized clinical trial. Endoscopy. 2016 Sep;48(9):823-8. doi: 10.1055/s-0042-108433. Epub 2016 Jun 15. PMID 27305424